CLINICAL TRIAL: NCT01916408
Title: The Effects of Oral Proteolytic and Hydrolytic Enzymes and Flavonoids on Inflammatory Markers and Coagulation After Marathon Running
Brief Title: The Effects of Enzymes and Flavonoids on Inflammation and Coagulation After Marathon
Acronym: Enzy-MagIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Enzy-MaGIC2013/1; 2013-001233-40 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-08-05 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Inflammation; Death, Sudden, Cardiac; Death; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Death, Sudden; Blood Coagulation Disorders; Respiratory Tract Infections
Keywords: Exercise; Inflammation; Upper Respiratory Tract Illness; Oral Proteolytic and Hydrolytic Enzymes; Flavinoids
MeSH Terms: conditions — Inflammation; Death, Sudden, Cardiac; Death; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Death, Sudden; Blood Coagulation Disorders; Respiratory Tract Infections; Motor Activity | interventions — Wobenzym

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wobenzym plus (Active Comparator): 3 x 4 tablets of the study medication each day for the one week before and 3 x 2 tablets of the study medication each day for the two weeks after the marathon.
  Interventions: Drug: Wobenzym plus
- Placebo PL1 (Placebo Comparator): 3 x 4 tablets of the study medication each day for the one week before and 3 x 2 tablets of the study medication each day for the two weeks after the marathon.
  Interventions: Drug: PL 1

INTERVENTIONS:
Drug: Wobenzym plus — 3 x 4 tablets of the study medication each day for the one week before and 3 x 2 tablets of the study medication each day for the two weeks after the marathon.
  Other Names: manufacturing authorisation number DE_BE_01_MIA_2012_0034/5373/1 - MUCOS/4
  Arms: Wobenzym plus
Drug: PL 1 — 3 x 4 tablets of the study medication each day for the one week before and 3 x 2 tablets of the study medication each day for the two weeks after the marathon.
  Other Names: Placebo
  Arms: Placebo PL1

SUMMARY:
The aim of the present study is to investigate changes in inflammatory status and incidence of infection after extreme aerobic physical stress (participation in a marathon). In addition, the impact of marathon running on the hemostasis and muscular state will be evaluated. Changes at the inflammatory, muscular, and rheological level will be related to ingestion of oral hydrolytic enzymes and bioflavonoids.

DETAILED DESCRIPTION:
The influence of extreme physical stress, such as that experienced during marathon competition, on the inflammatory system and coagulation has been investigated. However, up until now, countermeasures against these adverse effects are not adequately identified.

Immune-modulators (e.g. flavonoids) are known to be present in fruits and vegetables. There are also several different proteolytic and hydrolytic enzymes found in fruits most of whom are attributed protective properties. Therefore, 160 trained and untrained runners will consume a mixture of different enzymes and flavonoids (Wobenzym Plus®) or PL 1 (placebo) and effects on changes in inflammation and hemostasiologic parameters will be investigated during and after extreme physical stress (participation in a marathon race). The clinical result of the perturbation of the immune system will be assessed by the Wisconsin Upper Respiratory Symptom Survey (WURSS-24) with regard to symptoms of the upper respiratory tract system.

It is hypothesized that the intake of a product with immunomodulatory potential (Wobenzym Plus ®, consisting of hydrolytic enzymes and flavonoids) can positively influence both inflammation and blood coagulation pertubations observed after a marathon race.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male
* Age 20-65 years
* History of at least one successfully finished half marathon
* Intention to participate at the Munich Marathon 2013
* Subject is able to read, understand, and sign a written Informed Consent to participate in the Enzy-MagIC-Study

Exclusion Criteria:

* Known cardiac disease
* Known allergy against the active ingredient of the study medication or pineapple, papaya, or kiwi
* Known severe coagulopathy
* Known lactose intolerance
* Pharmaceutical treatment for diabetes mellitus or arterial hypertension
* Acute or chronic renal failure
* Acute or chronic liver disease
* Acute or chronic infection or inflammatory disease
* Use of medications or supplements influencing immune function
* Musculoskeletal or psychiatric disease
* Neoplasia
* Participation in other interventional trials

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The Effects of Oral Proteolytic and Hydrolytic Enzymes and Flavonoids on Inflammatory Markers after Marathon Running | one months
  Change of the inflammatory marker (IL-6) before and after a marathon in relation to the consumption of oral hydrolytic enzymes and bioflavonoids.

SECONDARY OUTCOMES:
The Effects of Oral Proteolytic and Hydrolytic Enzymes and Flavonoids on upper respiratory tract infections after Marathon Running | one months
  frequency of upper respiratory tract infections (URTI) post-marathon measured by WURSS-24 questionnaire before and after the marathon
The Effects of Oral Proteolytic and Hydrolytic Enzymes and Flavonoids on Coagulation after Marathon Running | 1 month
  changes in rheological parameters (platelets,tissue plasminogen activator (tPA), plasminogen activator inhibitor (PAI-1), aggregation time)
The Effects of Oral Proteolytic and Hydrolytic Enzymes and Flavonoids on muscular strain after Marathon Running | 1 month
  changes in muscular (CK, myoglobin)and muscular strain (McGill questionnaire)

OTHER OUTCOMES:
The Effects of Marathon Running on cardiac biomarkers | one months
  Controlling for cardiac biomarker (Hs-Troponin T, Hs-CRP, BNP)after marathon

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Scherr, Dr. med., Principal Investigator — Klinikum rechts der Isar der TUM
Locations (1):
- Department of Preventive and Rehabilitative Sports Medicine, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Scherr J, Halle M. Amendment on the findings of two previously published articles. Eur J Prev Cardiol. 2018 Mar;25(5):558. doi: 10.1177/2047487317754279. Epub 2018 Jan 26. No abstract available. PMID 29370708
- [Derived] Grabs V, Peres T, Zelger O, Haller B, Pressler A, Braun S, Halle M, Scherr J. Decreased prevalence of cardiac arrhythmias during and after vigorous and prolonged exercise in healthy male marathon runners. Am Heart J. 2015 Jul;170(1):149-55. doi: 10.1016/j.ahj.2015.04.001. Epub 2015 Apr 9. PMID 26093876
- [Derived] Grabs V, Nieman DC, Haller B, Halle M, Scherr J. The effects of oral hydrolytic enzymes and flavonoids on inflammatory markers and coagulation after marathon running: study protocol for a randomized, double-blind, placebo-controlled trial. BMC Sports Sci Med Rehabil. 2014 Feb 22;6(1):8. doi: 10.1186/2052-1847-6-8. PMID 24559067